CLINICAL TRIAL: NCT02207140
Title: Effect of Multi-species Probiotic HOWARU® Restore, on Gut Microbiota of Elderly
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Gabriella C. van Zanten (Other)
Responsible Party: Sponsor-Investigator, Gabriella C. van Zanten, Postdoc, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: DKID H-1-2014-051; H-1-2014-051 (Other: The Scientific Ethics Committee of the Capital Region, Denmark)
Record Dates: First submitted 2014-07-31; First posted 2014-08-04 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Elderly; Probiotics; Clostridium Difficile; Gut Microbiota; Fecal Metabolome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- probiotic (Experimental): HOWARU Restore
  Interventions: Dietary Supplement: HOWARU Restore
- placebo (Placebo Comparator): microcrystalline cellulose
  Interventions: Dietary Supplement: HOWARU Restore

INTERVENTIONS:
Dietary Supplement: HOWARU Restore

SUMMARY:
The study is randomized, double-blinded and placebo-controlled with a duration of 24 weeks. Following randomization, healthy elderly are randomized into two groups receiving probiotics or placebo. Fecal samples are collected before and after the study. The samples are investigated for Clostridium difficile levels, changes in diversity of the gut microbiota as well changes in the fecal metabolome. The effects of the produced metabolites on mitochondrial activity will moreover be investigated using selected intestinal cell lines.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* aged 75 years or more

Exclusion Criteria:

* Individuals with chronic bowel diseases
* Individuals with severe immunosuppression
* Individuals with dementia
* Individuals who are terminally ill
* If severe/prolonged illness occurs after the start of the test, the subject must drop out of the study
* Individuals who have consumed probiotic products after two weeks prior to the start of the study or during it.
* Subjects with a history of substance abuse
* Subjects that, in the investigators opinion, are not expected to complete the study succesfully

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Fecal Clostridium difficile numbers | 24 weeks

SECONDARY OUTCOMES:
fecal microbial composition | 24 weeks

OTHER OUTCOMES:
fecal metabolome | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella C van Zanten, PhD, Principal Investigator — University of Copenhagen, Dept. of Food Science
Locations (1):
- Department of Food Science, Food Microbiology, Faculty of Science, University of Copenhagen, Frederiksberg C, Denmark